CLINICAL TRIAL: NCT00367159
Title: Evaluation of the Efficiency of Autologous Adipocytes Graft in Endoscopic Treatment in Vesico-Renal Reflux in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Direction de la Recherche Clinique et de l'Innovation - Hôpitaux Universitaires de Strasbourg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3490; TC 197
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Vesico-Ureteral Reflux
Keywords: Vesico-ureteral reflux, autologous adipocytes, adipocytes graft
MeSH Terms: conditions — Vesico-Ureteral Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: endoscopic treatment of vesico-renal reflux — Autologous Adipocytes Graft (lipostructure)

SUMMARY:
Urinary tract infection (UTI) is a common problem in childhood associated with vesico-renal reflux (VRR) in 25-40% of children. A persistent VRR and repeated pyelonephritis may predispose to renal scarring and chronic renal failure with an end-stage renal failure in up to 3% of children.Defining a standard behaviour facing VRR in children is not easy because of the lack of reliable evidence. Numbers of studies compare prospectively or retrospectively, medical, endoscopical and surgical treatment.Surgical techniques are effective but invasive and not free of complication. Medical treatment is submissive to a good observance. The introduction of endoscopic techniques permits to prevent UTI and new renal failure by VRR elimination. Since the beginning of the endoscopic treatment, several bulking agents have been proposed. The ideal agent should be easy to inject, stable in time and should be safe. Of course it should be at least as efficient as actual bulking agent. The use of Teflon was the first wave of success of endoscopic treatment. But sudden passion of Teflon has been darkened by the notion of migration. Since, others substances have been proposed, autologous or exogenous, resorbable or not. But none was ideal and no solutions were found facing problem of biocompatibility or long-term stability.Using adipose tissue as a bulking agent is ancient in plastic surgery and indications had known a leap forward in the last century with Coleman who introduced a new technique called "lipostructure". This technique has known a growing interest in the restoration of all volume defects in plastic surgery because of the stability of the graft. We propose to apply this technique to VRR management in children in order to combine innocuousness and efficiency.

ELIGIBILITY:
Inclusion criteria :

* sexe : male and female
* age : 3 to 15 years
* written consent
* Vesico-renal reflux staged I to III revealed by a pyelonephritis ; after failure of medical treatment or parent refusal of medical treatment or initial renal failure.

Exclusion criteria :

* Before 3 years or older than 15 years
* insulino-dépendant diabet
* neurologic bladder
* abnormalities of the urinary tract
* kidney transplantation
* past history of bladder surgery
* anorexia (BMI <12)
* Vesico-renal reflux staged IV or V
* Active urinary tract infection

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2007-01; Primary Completion 2020-08 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Realization of an urethrocystography | at 3 months and 1 year

SECONDARY OUTCOMES:
Clinical or biological diagnosis of a pyelonephritis during the follow up (10 years) | Day 1; Month 1; Month 3 ; Year 1; Year 5 and Year 10

CONTACTS AND LOCATIONS:
Overall Officials: François BECMEUR, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Chirurgie Infantile, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg, France